CLINICAL TRIAL: NCT00154349
Title: Phase II Study of Imatinib Mesylate for Philadelphia-Positive Acute Lymphocytic Leukemia
Brief Title: Efficacy Study of Imatinib Mesylate to Treat Philadelphia-Positive Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571I1203
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphocytic Leukemia
Keywords: Ph+ALL; imatinib mesylate
MeSH Terms: interventions — Imatinib Mesylate

ARMS (1):
- imatinib mesylate (Experimental)
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate
  Other Names: STI571,; Glivec,; Gleevec

SUMMARY:
The objective of this study is to determine the efficacy and safety of imatinib mesylate in patients diagnosed as having Philadelphia chromosome positive acute lymphocytic leukemia (ALL).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of ALL.
* Patients confirmed to be Ph chromosome positive or bcr-abl gene positive.
* Patients in relapse
* Patients refractory to initial remission induction therapy
* Patients ineligible for initial remission induction therapy
* Patients with an ECOG Performance Status Score from 0 to 2
* Serum creatinine concentration of not more than 2 × the upper limit of the normal range (ULN)
* AST (SGOT) and ALT (SGPT) of not more than 3 × ULN. In patients with hepatic dysfunction from leukemic involvement, AST (SGOT) and ALT (SGPT) should be not more than 5 × ULN
* Serum bilirubin level not more than 3 × ULN

Exclusion Criteria:

* Patients with findings indicative of leukemic involvement of the central nervous system
* Patients with any serious concomitant medical condition (e.g., poorly controllable infection, interstitial pneumonia, pulmonary fibrosis, congestive cardiac failure, poorly controlled diabetes mellitus, mental disorder)
* Patients expected to receive any hematopoietic stem cell transplantation within 6 weeks of the planned initiation of the study drug
* Patients having received any hematopoietic stem cell transplantation who have a Grade 3 or 4 GVHD.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-10; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
3 month hematological response rate

SECONDARY OUTCOMES:
Duration of hematological response
Survival
Cytogenetic response in every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals